CLINICAL TRIAL: NCT00971828
Title: A Case-control Study to Assess Risk of Coronary Heart Disease in Idiopathic Inflammatory Myopathy
Status: Completed | Type: Observational
Sponsor: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Chinoy-001
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Idiopathic Inflammatory Myopathy
Keywords: Myositis; polymyositis; dermatomyositis
MeSH Terms: conditions — Myositis; Polymyositis; Dermatomyositis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bloods, including fasting blood sugar, lipid profile and C-reactive protein, serum creatine kinase, erythrocyte sedimentation rate, serology including antiphospholipid status.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Idiopathic inflammatory myopathy: IIM patients will be recruited via the Adult Onset Myositis clinic, Salford Royal NHS Foundation Trust. Suitable patients will be asked if they are willing to partake in the study, via a letter, including a patient information leaflet. If willing, they will contact our study co-ordinator, who will facilitate the visit to the WTCRF. The patient will then sign a consent form and be able to enter the study.

SUMMARY:
This study will be co-ordinated by Dr Hector Chinoy, Dr Robert G Cooper (Salford Royal NHS Foundation Trust / The University of Manchester) and Dr Ian N Bruce (Central Manchester University Hospitals NHS Foundation Trust/ The University of Manchester). An initial pilot study will be completed, to establish proof of concept of the study and to examine whether trends may observed of differences between cases and controls.

Twenty five prevalent UK Caucasian adult IIM cases, confirmed by internationally accepted criteria, will be recruited via the Adult Onset Myositis clinic, Salford Royal NHS Foundation Trust. Age, gender and race-matched controls will be recruited on a 'best friend' system. At the Wellcome Trust Clinical Research Facility (WTCRF), The University of Manchester, facilities are already available for B-mode ultrasound CIMT measurement, Endo-PAT, lean body mass measurement and contrast echocardiography. Cases and controls will have their cardiovascular risk factors assessed using a standardised questionnaire and blood tests. Further tests performed will include blood pressure, electrocardiogram, lean body mass, B-mode ultrasound CIMT measurement and Endo-PAT. IIM cases will have additional blood tests and a clinical assessment to assess their disease status, and contrast echocardiography. As part of a linked study, subjects (but not controls) will also have Gd-DTPA-MRI of the heart performed.

DETAILED DESCRIPTION:
This study will be coordinated by Dr Hector Chinoy, Dr Robert G Cooper (Salford Royal NHS Foundation Trust / The University of Manchester) and Dr Ian N Bruce (Central Manchester University Hospitals NHS Foundation Trust/ The University of Manchester). An initial pilot study will be completed, to establish proof of concept of the study and to examine whether trends may be observed of differences between cases and controls.

Thirty UK Caucasian adult IIM cases, confimed by internationally accepted criteria, will be recruited via the Adult Onset Myositis clinic, Salford Royal NHS Foundation Trust. Age, gender and racematched controls will be recruited on a 'best friend' system. STUDY METHODS:In order to establish whether CHD risk is increased in patients with myositis, we would like to perform a pilot study, comparing the cardiovascular risk factors of 30 patient's from Salford Royal's adult myositis clinic, with a group of 30 healthy controls. Participant would be invited along to the Wellcome Trust Clinical Research Facility (WTCRF), where all the necessary tests would be performed at a 'one off' study visit. Participants would be asked to bring along a friend of the same gender and roughly the same age, who would then comprise the 'healthy control' comparison group.

The study would involve a consultant clinician completing a 'heart disease questionnaire' for each of the participants.

A single blood sample would be taken to check their blood sugar levels and cholesterol, and if they had myositis, disease activity would also be assessed. The non invasive diagnostic testing would include an ultrasound of the blood vessels of the neck, checking for narrowing of the arteries, and a special blood pressure test, looking for the early signs of atherosclerosis (build up of fat in the blood vessels). An electrocardiogram (ECG) would be performed, and if they have myositis, an ultrasound test of their heart (echocardiogram), would also be performed. A gadoliniumenhanced magnetic resonance scan (GdDTPAMRI) of the heart will be performed to examine for inflammation of the heart tissue (pericardium and myocardium). The echo and MR will only be performed in patients, and not controls.

If the study demonstrated that patients with myositis had more chance of developing CHD, than those in the control group, this would have implications for their future clinical care, requiring close monitoring of patients for the early signs of CHD, and the appropriate intervention when necessary. This study will be funded by the WTCRF Small Grants Award Scheme.MORE DETAILED DESCRIPTION OF STUDY METHODS:Cases and controls will have the following recorded for assessment of cardiovascular risk factors: i) Standardised questionnaire to ascertain basic details, e.g. age, ethnicity, medical and family history, drug use and smoking. ii) Height and weight measurement. iii) Blood tests, including fasting blood sugar, lipid profile & Creactive protein. iv) Lean body mass measurement using a body composition analyser. v) Electrocardiogram. v) Subclinical atherosclerosis measurement using Bmode ultrasound CIMT. vi) Endothelial dysfunction measurement using EndoPAT.

Cases will additionally have the following to assess disease status:

i) Clinical assessment of myositis disease activity (MITAX/MYOACT) and disease damage (MDI, MYODAM). ii) Assessment of muscle strength using manual muscle testing. iii) Further bloods including serum creatine kinase, erythrocyte sedimentation rate, serology including antiphospholipid status. iv) Assessment of left ventricular/septal dysfunction, and pericardial abnormalities using contrast echocardiography. vi) Assessment of the diagnostic utility of GdDTPAMRI to assess myocardial disease activity in the presence of cardiovascular disease. All procedures will be conducted by a technician or nurse employed within the WTCRF. The clinical and muscle strength assessment will be performed by a medical practitioner (to be appointed).

At the WTCRF, The University of Manchester, facilities are already available for Bmode ultrasound CIMT measurement, EndoPAT, lean body mass measurement and contrast echocardiography. Cases and controls will have their cardiovascular risk factors assessed using a standardised questionnaire and blood tests. Further tests performed will include blood pressure, electrocardiogram, lean body mass, Bmode ultrasound carotid artery narrowing and EndoPAT. IIM cases will have additional blood tests and a clinical assessment to assess their disease status. As part of a linked study, subjects (but not controls) will also have GdDTPAMRI and contrast echocardiography of the heart performed. The primary research end point will be the detection of significant patient/control group differences.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be age, sex and race matched and willing to take part in the study.

Exclusion Criteria:

* Any subject below the age of 18 years, or
* Any subject with a personal or family history of past or current inflammatory or connective tissue diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IIM patients will be recruited via the Adult Onset Myositis clinic, Salford Royal NHS Foundation Trust. Suitable patients will be asked if they are willing to partake in the study, via a letter, including a patient information leaflet. If willing, they will contact our study co-ordinator, who will facilitate the visit to the WTCRF. The patient will then sign a consent form and be able to enter the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hector Chinoy, PhD MRCP, Principal Investigator — Northern Care Alliance NHS Foundation Trust
Locations (1):
- Welcome Trust Clinical Research Facility, Manchester, United Kingdom